CLINICAL TRIAL: NCT07178756
Title: ACUPUNCTURE FOR THE POSTOPERATIVE RECOVERY OF HIP FRACTURE PATIENTS: A PILOT RANDOMIZED CONTROLLED TRIAL
Acronym: AFTPROHFP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Khoo Teck Puat Hospital (Other)
Collaborators: Ministry of Health, Singapore (Other Government)
Responsible Party: Principal Investigator, Ong Zhi Lin Melissa, Dr Antony Xavier Rex Premchand, Senior Consultant; Specialties/Sub-Specialties Orthopaedic Surgery, Khoo Teck Puat Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019/01168
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Hip Fracture Surgeries; Post-operative Hip Fractures Recovery
Keywords: Acupuncture; Hip fracture surgery; Post hip fracture surgery recovery; Hip fracture
MeSH Terms: conditions — Hip Fractures | interventions — Acupuncture Therapy; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Randomization: Patients will be randomized to either Group A, where they receive postoperative management AND acupuncture, or Group B, where they receive postoperative management ONLY. Acupuncture will be performed on patients in Group (A) 2x/week from POW 5 to POW 8, a total of 8 acupuncture treatments will be administered. From the 2nd to 8th treatment, electroacupuncture and infrared therapeutic lamp will be used.
  The acupuncture needles used for this study are Kinhong/MAC sterile acupuncture needles for single use. The depth of needle insertion will range from 1-1.5cm and needles will be left in situ for 20 minutes. The following acupuncture points will be used bilaterally for this study: 1) Li 4 (Hegu), 2) St 36 (Zusanli) , 3) Sp 6 (Sanyinjiao), 4) Sp 9 (Yinlingquan), 5) Sp 10 (Xuehai), 6) Kd 3 (Taixi) 7) Gb 34 (Yanglinquan), 8) Ren 6 (Qihai), 9), Auricular point - Kuan 10) Auricular point - Shen Men
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization/Allocation Concealment: 1) KTPH CRU Biostatistician (non-study team member) will use a random number generator to create a random sequence for the subjects. There will be a corresponding subject number in running sequence to each randomized generated number. The randomized numbers will then be categorized into 2 groups, odd numbers into either acupuncture or control group then even numbers into the other. 2) 90 opaque sealed envelopes will be prepared for 90 subjects. The subject number will be written on the front of each envelope. Inside each envelope, there is an insert stating the group which the subject is allocated to. 3) These sealed envelopes will be handed over to the study team. The study team member will take the relevant envelope in accordance with the subject number to check what group the subject is allocated to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture Group (Group A) (Experimental): In addition to standard postoperative management program, acupuncture treatment will be added
  Interventions: Procedure: Acupuncture
- Control Group (Group B) (Other): Only receive standard postoperative management which includes: conventional analgesia and physiotherapy. No acupuncture given
  Interventions: Other: Post-operative standard care

INTERVENTIONS:
Procedure: Acupuncture — Both groups A and B will undergo standard postoperative management program. This includes conventional analgesia and physiotherapy POD 1, 2 and 3, followed by 5x/week until discharge, post-discharge, patients will continue physiotherapy 1-2x/ week for 3 months depending on their rate of recovery.
  In addition, acupuncture treatment will be delivered for the treatment group. Acupuncture will be performed 2x/week from postoperative week (POW) 5 to POW 8, a total of 8 acupuncture treatments will be administered. From the 2nd to 8th treatment, electroacupuncture and infrared therapeutic lamp will be used. The acupuncture needles to be used for this study are Kinhong/MAC sterile acupuncture needles for single use. The needles will be left in situ for 20 minutes. Electrical stimulation will be delivered at 2Hz for 20 min, at an intensity below individual patient's pain threshold. 4 acupuncture points will be stimulated in pairs.
  Other Names: Acupuncture in addition to standard care; Acupuncture AND physiotherapy; Acupuncture in addition to standard post operative management for hip fracture patients
  Arms: Acupuncture Group (Group A)
Other: Post-operative standard care — Standard postoperative management program includes: conventional analgesia and physiotherapy POD 1, 2 and 3, followed by 5x/week until discharge. Post-discharge, patients will continue physiotherapy 1-2x/ week for 3 months depending on their rate of recovery. No acupuncture given
  Other Names: Standard post-operative management program for hip fracture
  Arms: Control Group (Group B)

SUMMARY:
Hip surgery is a common and safe medical intervention to restore the functionality and mobility of the hip joint in patients suffering from hip fractures. Despite the advances in surgical techniques, a relatively large proportion of patients suffer from postoperative pain, joint dysfunction and loss of muscle strength. These outcomes hinder rehabilitation, which consequently imposes significant economic burden for health systems.

This study aims to assess if the addition of acupuncture to existing postoperative management will improve the following patient outcomes post hip surgery:

1. Postoperative pain
2. Function (muscular strength and mobility)

Methods Patients who underwent hip surgery due to unilateral hip fracture, who fulfill the inclusion and exclusion criteria, will be randomly allocated to either receive postoperative management ONLY (Conventional analgesics and physiotherapy) or with the addition of acupuncture post hip surgery.

In additional to standard care, acupuncture will be performed on patients in Group A twice a week from post-operative week (POW) 5 to 8, a total of 8 acupuncture treatments will be administered. From the 2nd to 8th treatment, electroacupuncture and infrared therapeutic lamp will be used. Group B will receive only standard post-operative management.

For patients in both Group A and B, primary outcomes will be assessed at the following time points: Post- Operative Week (POW) 0, 6, Post-Operative Month (POM) 6 and 12, while the secondary outcomes will be assessed at the following time points: POW 6, POM 6 and 12. The Primary Outcomes include:1. Modified Harris Hip Score 2. Visual Analogue Scale (VAS-100). The Secondary Outcomes include: 1. Timed Up and Go (TUG) assessment. The TUG assessment will be performed thrice during each assessment and an average time will be taken. 2. Lower extremity muscle strength measured using a portable dynamometer. The subject's operated and non-operated side will be measured.

Hypothesis The addition of acupuncture to existing postoperative management will reduce pain and enhance functional recovery, better and faster than with postoperative management alone.

ELIGIBILITY:
Inclusion Criteria:

Patients who undergone surgery due to unilateral hip fracture. Patients aged 40-99 (male), 55-99 (female). Ambulatory with or without aid prior to hip fracture. Able provide consent for the study and acupuncture treatment. Able to attend all treatment sessions

Exclusion Criteria:

Patients with morbid obesity (Body Mass Index >40) . Patients with communication barriers such as aphasia or language . Local or systemic infection or dermatological disease affecting sites of acupuncture. Existing treatment with anti-neoplastic, oral corticoid or immunosuppressive drugs. Needle phobia or inability to stay still for 30 min during acupuncture retention . History of psychiatric disease, kidney failure on peritoneal dialysis, substance abuse . If there exist any postoperative complications that deviate from standard management, resulting in interference of patient's clinical evaluation

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-10-21 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-11-14 (Estimated)

PRIMARY OUTCOMES:
1. Modified Harris Hip Score | postoperative Week (POW) 0, 6, postoperative month (POM) 6 and POM 12
  Assessing pain and function
Visual Analogue Scale (VAS)-100 | postoperative Week (POW) 0, 6, postoperative month (POM) 6 and POM 12
  For assessing the pain intensity

SECONDARY OUTCOMES:
Timed get Up and Go (TUG) test | POW 6, POM 6 and 12
  Test for assessing function (Gait and speed). The TUG will be performed thrice during each assessment and the average time will be taken.
Lower extremity muscle strength | POW 6, POM 6 and 12
  Lower extremity muscle strength will be measured using a portable dynamometer. The subject's operated and non-operated side will be measured.

CONTACTS AND LOCATIONS:
Locations (2):
- Singapore (2):
  - Admiralty Medical Centre (Khoo Teck Puat Hospital- KTPH @ ADMC ), Singapore
  - Khoo Teck Puat Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seitz DP, Anderson GM, Austin PC, Gruneir A, Gill SS, Bell CM, Rochon PA. Effects of impairment in activities of daily living on predicting mortality following hip fracture surgery in studies using administrative healthcare databases. BMC Geriatr. 2014 Jan 28;14:9. doi: 10.1186/1471-2318-14-9. PMID 24472282
- [Background] Chan MWC, Wu XY, Wu JCY, Wong SYS, Chung VCH. Safety of Acupuncture: Overview of Systematic Reviews. Sci Rep. 2017 Jun 13;7(1):3369. doi: 10.1038/s41598-017-03272-0. PMID 28611366
- [Background] Usichenko TI, Dinse M, Hermsen M, Witstruck T, Pavlovic D, Lehmann C. Auricular acupuncture for pain relief after total hip arthroplasty - a randomized controlled study. Pain. 2005 Apr;114(3):320-327. doi: 10.1016/j.pain.2004.08.021. PMID 15777857
- [Background] Mikashima Y, Takagi T, Tomatsu T, Horikoshi M, Ikari K, Momohara S. Efficacy of acupuncture during post-acute phase of rehabilitation after total knee arthroplasty. J Tradit Chin Med. 2012 Dec;32(4):545-8. doi: 10.1016/s0254-6272(13)60068-0. PMID 23427386

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-02): https://cdn.clinicaltrials.gov/large-docs/56/NCT07178756/Prot_SAP_000.pdf